CLINICAL TRIAL: NCT05109117
Title: A Clinical Study to Evaluate the 8-Hour Moisturization Efficacy of an Over-The-Counter Sunscreen Lip Balm After a Single Application
Brief Title: Clinical Study to Evaluate the Efficacy of an Over-the-counter (OTC) Sunscreen Lip Balm Product
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HALEON (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 218006
Record Dates: First submitted 2021-10-26; First posted 2021-11-05 (Actual); Results first posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2023-10

CONDITIONS: Sunscreening Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test Arm (Experimental): Single topical application: 80 +/- 2 milligrams (mg) (2.0 +/- 0.05 mg/centimeter^2) of ChapStick Active Performance (CAP) Unscented will be applied to the assigned test site using a fingercot. The test product will be evenly spread over the test site using light pressure.
  Interventions: Drug: CAP Unscented
- Control Arm (No Intervention): No treatment will be applied to the assigned control site.

INTERVENTIONS:
Drug: CAP Unscented — Sunscreen lip balm.
  Arms: Test Arm

SUMMARY:
The purpose of this study is to evaluate the 8-hour moisturization efficacy of OTC sunscreen lip balm after a single treatment application.

DETAILED DESCRIPTION:
A single-center, randomized, controlled, intra-individual comparison, open label clinical study to determine the 8-hour moisturization efficacy of a sunscreen lip balm. Skin hydration will be assessed before (Baseline) and after (2, 4, 6 and 8 hours post-treatment) a single treatment with test product, compared to 'no treatment' as control, using a corneometer. Study treatments will be randomly assigned to 2 test sites delineated on the skin of the participant's volar forearms (one test site on each arm). A 1-week conditioning phase will precede the test day, during which participants will use the soap provided for personal washing.

ELIGIBILITY:
Inclusion Criteria:

* Participant must provide a signed and dated, legally effective, informed consent document, which indicates they have been informed of, and understand, all pertinent aspects of the study, before any study procedures are performed (in conformance with 21 Code of Federal Regulations [CFR] Part 50: 'Protection of Human Subjects.')
* Participant must provide relevant details of their medical history and current/recent medications and treatments.
* Participant has completed a Health Insurance Portability and Accountability Act (HIPAA) Authorization Form in conformance with 45 CFR Parts 160 and 164.
* Participant must have completed a Photo Release Form.
* Participant must be able to read, write, speak and understand English.
* Participant must be in good general health.
* Participant must have a valid form of personal identification (photo identity [ID], driver's license, passport, permanent resident card, military ID card; forms cannot be expired)
* Male and female participants of child-bearing potential must agree to use a highly effective method of contraception for the duration of the study and for 14 days after treatment application. (Note: A participant is considered to be of child-bearing potential if, in the opinion of the Principle investigator [PI], they are biologically capable of having children and sexually active.
* Participant must agree to be sequestered in a temperature/humidity monitored test room at the clinical site (temperature 21 degree Celsius [C] +/- 2 degree C, relative humidity [RH] 50 percent [%] +/- 10%) for the duration of the test day (Visit 2), approximately 9.5 hours.
* Participant must agree to bring their own food (dry) and beverages to be consumed on the test day (Visit 2).
* Participant must agree not to consume hot or very cold food/beverages on the test day (Visit 2).
* Participant must agree to use the non-moisturizing soap provided for all personal washing during the conditioning phase of the study.
* Participant must agree to wear loose clothing for ease of access to the test sites (arms) and/or sleeves that can be easily rolled up.
* Participant must agree not to introduce any new cosmetic/toiletry products into their personal care regimen during the study.
* Participant must agree to refrain from any physical effort which might result in thermal regulation by sweating (for example, exercise class, rapid climbing of flights of stairs, jogging, cycling, brisk walking) for at least 2 hours prior to arriving the test day (Visit 2).
* Participant must agree to refrain from prolonged or excessive ultraviolet (UV) exposure (for example, sunbathing, tanning beds) for the duration of the study.
* Participant should be dependable and able to follow directions as outlined in the protocol and Informed Consent Form (ICF).

Exclusion Criteria:

* Participant with scheduled or planned Covid-19 vaccination during likely dates of study participation.
* Female participant who is pregnant, planning to become pregnant during the study, or breastfeeding ( self-reported).
* Participant with a history of sensitivity to any ingredient of the test material or skin marker pen, or latex; or any known sensitivities/allergies, including but not limited to cosmetic/toiletry products and topically applied skin treatment products/drugs.
* Participant with a history of an acute or chronic dermatologic, medical and/or physical condition that would, in the opinion of the investigator, confound study outcomes or increase the risk associated with participation. (Note: dry skin is not an exclusion per se; however, a participant with a level of dryness on the skin of the volar forearms that would, in the opinion of the investigator, confound study outcomes or increase the risk associated with participation should be excluded.
* Participant with a history of skin cancer, or currently undergoing treatment for active cancer of any kind.
* Participant with diabetes.
* Participant with a planned medical treatment/vaccination (other than the Covid-19 vaccination) during the study that would, in the opinion of the investigator, confound study outcomes or increase the risk associated with participation.
* Participant with a planned hospitalization during the study.
* Participant who is currently using, or has used in the past week, any systemic or topical corticosteroid, non-steroid anti-inflammatory drug, antihistamine, sympathomimetic, and/or vasoconstrictor or any other medication that would, in the opinion of the investigator, confound study outcomes or increase the risk associated with participation.
* Participant who is unwilling to cease use of personal care products (for example, moisturizers, lotions, sunscreens, sunless tanners) and/or topical medications at the test sites for the duration of the study.
* Participant who has had extensive UV exposure within 3 weeks of Screening (Visit 1).
* Participant with visual signs of irritation, sunburn, rashes, scratches, burn marks, scarring at the test sites that would interfere with corneometry measurements.
* Participant with excessive hair at the test sites that would interfere with corneometry measurements.
* Participant who has participated in a study involving the arms as a test site, or any other type of clinical study, within three weeks of screening (Visit 1).
* Participant who is an employee/contractor or immediate family member of the PI, study site or Sponsor.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- GSK Investigational Site, Piscataway, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, ICF
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoint and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at single center in United States.
Pre-assignment Details: Two test sites on each participant's volar forearms (one site per arm) were randomized to treatment, either ChapStick Active Performance (CAP) Unscented (test product) or no treatment (control).
Units Other Than Participants: Volar forearm test sites
Groups:
- All Study Participants: Study participants were randomly assigned to receive a single topical application of CAP Unscented (test product) or no treatment (control) to two 40 square centimeter (cm^2) test sites delineated on the skin of their volar forearms. 80 +/- 2 milligrams (mg) CAP Unscented was applied to its assigned test site (2.00 +/- 0.05 mg/cm^2); no treatment was applied to the test site on the opposing volar forearm. Skin hydration was assessed using corneometry (3 readings per test site at each timepoint), the higher the corneometer reading, the more hydrated the skin.
Period: Overall Study
Arm/Group | All Study Participants
Started | 38; 76 Volar forearm test sites
Safety Population | 37; 74 Volar forearm test sites
Test Product (CAP UnScented) | 36; 36 Volar forearm test sites
Control (No Treatment) | 36; 36 Volar forearm test sites
Completed | 36; 72 Volar forearm test sites
Not Completed | 2; 4 Volar forearm test sites
Not completed — Lost to Follow-up | 1
Not completed — Discontinued for non-compliance | 1

BASELINE CHARACTERISTICS:
Population: Safety population: included all randomized participants who received study treatment.
Groups:
- All Study Participants: Study participants were randomly assigned to receive a single topical application of CAP Unscented (test product) or no treatment (control) to two 40 cm^2 test sites delineated on the skin of their volar forearms. 80 +/- 2 mg CAP Unscented was applied to its assigned test site (2.00 +/- 0.05 mg/cm^2); no treatment was applied to the test site on the opposing volar forearm. Skin hydration was assessed using corneometry (3 readings per test site at each timepoint), the higher the corneometer reading, the more hydrated the skin.
Arm/Group | All Study Participants
Number analyzed (Participants) | 37
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.6 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Corneometer Measurements
Description: Corneometry is an instrumental technique. It uses a capacitance sensor to measure the dielectric constant of the stratum corneum which is directly proportional to the water content of the skin (skin hydration). Capacitance of the skin surface is expressed in arbitrary units of skin hydration; the higher value, the more hydrated (moist) the skin. The mean of 3 corneometer readings taken for each test site at each assessment timepoint (Baseline and 2, 4, 6 and 8 hours post-treatment) was calculated for each individual participant. Change from Baseline was calculated at each post-treatment timepoint as the post-treatment value minus the Baseline value.
Time Frame: Baseline (pre-treatment), 2, 4, 6 and 8 hours post-treatment
Population: Primary analysis population: included all eligible participants who were randomized, received study treatment and provided at least one post-treatment efficacy assessment.
Measure: Mean (Standard Deviation); unit: Arbitrary units
Units Other Than Participants: Volar forearm test sites
Groups:
- Test Product: All participants who received CAP Unscented at the assigned test site and provided at least one post-treatment efficacy assessment.
- Control (No Treatment): All participants who received no treatment at the assigned test site and provided at least one post-treatment efficacy assessment.
Arm/Group | Test Product | Control (No Treatment)
Number analyzed (Participants) | 36 | 36
Number analyzed (Volar forearm test sites) | 36 | 36
Arbitrary units
  Baseline | 23.5 (5.7) | 24.2 (6.0)
  Change from Baseline 2 hours post-treatment | 2.4 (4.2) | -0.6 (2.3)
  Change from Baseline 4 hours post-treatment | 1.7 (3.5) | -0.1 (2.7)
  Change from Baseline 6 hours post-treatment | 2.0 (5.3) | 0.0 (2.6)
  Change from Baseline 8 hours post-treatment | 1.0 (3.3) | -0.2 (2.7)
Statistical Analysis 1: Comparison: Test Product vs Control (No Treatment); Pairwise comparison between Treated and Untreated sites 2 hours post-treatment; Test type: Superiority; p < 0.0001, ANCOVA; Analysis of Covariance (ANCOVA) model with treatment, timepoint, treatment*timepoint (interaction) and subject as terms; Baseline value as covariate; Adjusted Mean Difference = 2.8, 95% CI 2-sided [1.7 to 3.9]
Statistical Analysis 2: Comparison: Test Product vs Control (No Treatment); Pairwise comparison between Treated and Untreated sites 4 hours post-treatment; Test type: Superiority; p = 0.0077, ANCOVA; ANCOVA model with treatment, timepoint, treatment*timepoint (interaction) and subject as terms; Baseline value as covariate; Adjusted Mean Difference = 1.5, 95% CI 2-sided [0.4 to 2.7]
Statistical Analysis 3: Comparison: Test Product vs Control (No Treatment); Pairwise comparison between Treated and Untreated sites 6 hours post-treatment; Test type: Superiority; p = 0.0019, ANCOVA; [statistical method as in outcome 1, analysis 2]; Adjusted Mean Difference = 1.8, 95% CI 2-sided [0.7 to 2.9]
Statistical Analysis 4: Comparison: Test Product vs Control (No Treatment); Pairwise comparison between Treated and Untreated sites 8 hours post-treatment; Test type: Superiority; p = 0.0707, ANCOVA; [statistical method as in outcome 1, analysis 2]; Adjusted Mean Difference = 1.0, 95% CI 2-sided [-0.1 to 2.2]

2. Secondary Outcome: Percentage of Participants With Improved Corneometer Measurement
Description: Percentage of participants with improved corneometer measurement was calculated at each post-treatment timepoint as the number of participants who exhibited improvement (positive change) divided by the total number of participants included in the analysis.
Time Frame: 2, 4, 6 and 8 hours post-treatment
Population: Primary analysis population
Measure: Number; unit: Percentage of participant
Units Other Than Participants: Volar forearm test sites
Arm/Group | Test Product | Control (No Treatment)
Number analyzed (Participants) | 36 | 36
Number analyzed (Volar forearm test sites) | 36 | 36
Percentage of participant
  2 hours post-treatment | 69.4 | 38.9
  4 hours post-treatment | 66.7 | 44.4
  6 hours post-treatment | 66.7 | 55.6
  8 hours post-treatment | 66.7 | 50.0

ADVERSE EVENTS:
Time Frame: From screening until 14 days after last administration of study product (or last study procedure).
Description: Adverse events (AEs), and therefore all serious adverse events (SAEs), were to be collected from immediately after a participant provided written consent to participate in the trial until 14 days following the last administration of test material (or the last study procedure). All SAEs were to be reported within 24 hours of detection. AEs were to be classified by Intensity (mild, moderate, severe); Causality (probable, possible, unlikely); Seriousness (serious or non-serious).
Arm/Group | All Study Participants
All-Cause Mortality (participants affected / at risk) | 0/37
Serious Adverse Events (participants affected / at risk) | 0/37
Other Adverse Events (participants affected / at risk) | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
HALEON agreements may vary with individual investigators but will not prohibit any investigator from publishing. HALEON supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-28): https://cdn.clinicaltrials.gov/large-docs/17/NCT05109117/Prot_SAP_000.pdf